CLINICAL TRIAL: NCT07181655
Title: The Effectiveness of Intermittent Fasting, Caloric Restriction and Physical Activity Intervention On Metabolic Syndrome Biomarkers Among Adults With Metabolic Syndrome at Hospitals in Riyadh, Saudi Arabia
Brief Title: The Effectiveness of Intermittent Fasting, Caloric Restriction and Physical Activity On Metabolic Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, LAMIA SALEM A ALMAZID, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UPM-PhD LALMAZID
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; MetS
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Intermittent Fasting (Other): Intervention program of modified Intermittent fasting (Intermittent fasting, caloric restriction and physical activity)
  Interventions: Other: Modified Intermittent Fasting
- Control group: No Intervention (No Intervention): A control group receiving standard care provided by hospital

INTERVENTIONS:
Other: Modified Intermittent Fasting — Participants in Intervention group will follow a structured intermittent fasting protocol, specifically the 16:8 method, where they fast for 16 consecutive hours each day and restrict their eating to an 8-hour window. The fasting period can be personalized to suit individual schedules. During these fasting hours, participants must abstain from all foods and caloric drinks, but are encouraged to stay hydrated with non-caloric beverages and they will follow a structured, calorie-restricted diet, tailored to them, using a developed Food Frequency Questionnaire tool to select their daily calorie intake across sections to identify appropriate foods and beverages for patients with metabolic conditions. They will be prescribed to engage in at least 150 minutes per week of moderate intensity aerobic activities, such as brisk walking will be measured and evaluated using the mobile application of physical activity recommended by the Ministry of Health in Saudi Arabia.
  Other Names: Intervention Group
  Arms: Modified Intermittent Fasting

SUMMARY:
Metabolic syndrome (MetS) is a global health issue defined by a cluster of risk factors-abdominal obesity, elevated blood pressure, high fasting blood sugar, high triglycerides, and low HDL cholesterol-that together significantly increase the risk of cardiovascular disease, type 2 diabetes, and overall mortality. Globally, about 20-25% of adults are affected, but prevalence varies by region and population; in Saudi Arabia, studies report rates ranging from 28.3% to 56.4%, with higher rates observed in northern and central regions and among men. Major contributors to MetS in Saudi Arabia include obesity, sedentary lifestyle, smoking, and poor dietary habits, such as low fruit consumption. Effective management strategies focus on weight loss through caloric restriction, intermittent fasting, and increased physical activity, all of which have demonstrated improvements in metabolic markers like insulin sensitivity, blood pressure, and lipid profiles. Despite international evidence supporting these interventions, no randomized controlled trials have yet evaluated the combined effects of these approaches on MetS biomarkers in Saudi adults, underscoring the need for targeted research and public health initiatives to address the high and regionally variable burden of MetS in the country.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of interventions involving intermittent fasting, physical activity, and caloric restriction on metabolic syndrome biomarkers, body composition and lifestyle characteristics among patients with metabolic syndrome in Riyadh, Saudi Arabia. A randomized controlled trial (RCT) will be conducted at two hospitals, with 140 participants randomly assigned to two groups: Intervention Group the participants will be engaged in Intervention program of modified IF (Intermittent fasting, caloric restriction and physical activity) and Control Group: the participants will be engaged standard intervention provided by hospital. The primary outcomes will include changes in glycemic control (fasting blood glucose, HbA1c), cardiovascular risk markers (blood pressure, lipid profile), anthropometric measures (weight, BMI, waist circumference), physical activity levels, sleep quality, and dietary intake, assessed before and after the intervention to determine the comparative effectiveness of each approach on MetS biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria will be adult aged 18 years and above who have three or more of the following five risk factors (Kunduraci & Ozbek, 2020):

  * Abdominal obesity.
  * Elevated triglycerides.
  * Low HDL cholesterol.
  * Elevated blood pressure.
  * Elevated fasting blood glucose.

Exclusion Criteria:

* Being pregnant, lactating women.
* Diagnosis of cardiac failure or/and severe renal or liver diseases, cancer.
* Having had bariatric surgery.
* Physical or mental disability.
* Neurological or cognitive impairment.
* Participant with severely impaired vision, hearing, or speech.
* Following a special diet or having changed their dietary pattern within the previous 12 weeks of the study's start date.
* Use of insulin or sulphonamide derivative oral antidiabetic drugs.
* Conditions that will seriously affect weight management such as having had bariatric surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Blood Glucose Levels | Time Frame: Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 4 (4-week post 1 intervention). Timepoint 3 = week 8 (4-week post 2 intervention).Timepoint 4 = week 12 (12-week post 3 intervention
  Fasting plasma glucose and Random blood glucose will be measured using a spectrophotometer. The normal range of the Fasting plasma glucose is (5.6 - 6.9 mmol/l) and for Random blood glucose is (7.8-11.0 mmol/l).
Change in cholesterol Levels | Time Frame: Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 4 (4-week post 1 intervention). Timepoint 3 = week 8 (4-week post 2 intervention).Timepoint 4 = week 12 (12-week post 3 intervention
  Total cholesterol includes both High density lipoprotein cholesterol (HDL) and Low density lipoprotein cholesterol (LDL) will be measured using a spectrophotometer. The normal range of the total cholesterol is (≤ 5.2 mmol/l). While the normal range of LDL-cholesterol is (# 2.6 mmol/l) and HDL-cholesterol is (# 1.3 mmol/l)
Change in Blood Pressure | Time Frame: Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 4 (4-week post 1 intervention). Timepoint 3 = week 8 (4-week post 2 intervention).Timepoint 4 = week 12 (12-week post 3 intervention
  Blood pressure will be measured using sphygmomanometer. Normal blood pressure is usually considered to be between 120/80 mmHg.
Change the Body mass index (BMI) | Time Frame: Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 4 (4-week post 1 intervention). Timepoint 3 = week 8 (4-week post 2 intervention).Timepoint 4 = week 12 (12-week post 3 intervention
  The Body mass index (BMI) will be report in kg/m^2 by using the following formula (BMI = kg/m2 where kg is a
Change in physical activity | Time Frame: Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 4 (4-week post 1 intervention). Timepoint 3 = week 8 (4-week post 2 intervention).Timepoint 4 = week 12 (12-week post 3 intervention
  Physical activity will be assessed using the International Physical Activity Questionnaire (IPAQ), where time spent on various activity types was summed to determine weekly totals, and frequency, duration, and intensity were converted into metabolic equivalent (MET) values using standard tables
Change in dietary intakes | Time Frame: Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 4 (4-week post 1 intervention). Timepoint 3 = week 8 (4-week post 2 intervention).Timepoint 4 = week 12 (12-week post 3 intervention
  The dietary recall method will be implemented twice a week (Fridays and Mondays) to evaluate participants' food intake. The use of the FFQ of MetS (Phase 2) is essential as an effective intervention tool to support the health plan.two non-consecutive days (one usual day and one weekend day).

SECONDARY OUTCOMES:
Change in sleep quality | Time Frame: Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 4 (4-week post 1 intervention). Timepoint 3 = week 8 (4-week post 2 intervention).Timepoint 4 = week 12 (12-week post 3 intervention
  Participants' sleep quality will be evaluated using the Pittsburgh Sleep Quality Index (PSQI). The PSQI is the predominant method for measuring daytime sleepiness. Responses will be scored from 0 to 3, with the higher scores indicating acute sleep disturbances. asked to rate their chances of dozing during certain daily activities using ratings range from 0 (never doze) to 3 (high chance of dozing). Scores range from 0 to 24. An ESS score greater than 10 indicates excessive daytime sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Hazizi Abu Saad, PhD, Study Director — Universiti Putra Malaysia, 43400 Serdang, Selangor, Malaysia
Locations (1):
- Associate Professor Dr. Hazizi Abu Saad, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No